CLINICAL TRIAL: NCT06496711
Title: IMPLEMENT - Model Project for the Cross-sector Implementation of a Comprehensive and Quality-assured Sports and Exercise Therapy for Cancer Patients
Brief Title: IMPLEMENT - Model Project for Quality-assured Exercise Therapy for Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Leibniz Institute for Prevention Research and Epidemiology - BIPS GmbH (Other); University of Regensburg (Other); Ludwig-Maximilians - University of Munich (Other); Technical University of Munich (Other); Martin-Luther-Universität Halle-Wittenberg (Other); University Hospital Schleswig-Holstein (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Freerk Baumann; Prof. Dr., Prof. Dr. Freerk Baumann, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCologne 70114696
Record Dates: First submitted 2024-05-22; First posted 2024-07-11 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Cancer
Keywords: exercise therapy; Implementation
MeSH Terms: conditions — Neoplasms | interventions — Academies and Institutes

STUDY DESIGN:
Intervention Model Description: explorative, open, non-randomised mixed-methods study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer Patients and Parents of Cancer Patients (Other): Children: Age 5-12 years Parents of children with cancer Teenager: Age 13-17 years Parents of teenager with cancer AYAs: Adolescence and young adults: Age 18-39 years Adults: > 40 years
  Interventions: Other: Cancer Patients; Institutions and their employees in the treatment and/or counseling of cancer patients

INTERVENTIONS:
Other: Cancer Patients; Institutions and their employees in the treatment and/or counseling of cancer patients — The study population will be surveyed at 3 yearly measurement time points by means of questionnaires and interviews on attitudes, barrier and support factors for participation in exercise therapy.

SUMMARY:
IMPLEMENT aims to develop, test and establish a sustainable access structure for quality-assured oncological exercise therapy (qOET) in Germany as a model within the funding period of three years. This will be done in three phases:

Phase 1: In the first step, a characterization of the existing implementation structures and the existing barriers and needs as well as the establishment of the cooperation with the most important actors in the care system will take place.

Phase 2: In the subsequent implementation process, concrete measures are practically implemented in subprojects for specific target groups (children/adolescents, adults) and specific regions (rural, urban) as well as the digital solutions and interface management. With the help of a mixed-methods design, the barriers and facilitating factors of the implementation of area-wide qSBT will be investigated during the project and fed into a "learning system" for adaptation and improvement.

Phase 3: The success of the measures to increase patient participation in qOET and the development of the structures as well as the barrier and facilitating factors for an effective implementation will be addressed in a before-after comparison through evaluation steps and an economic accompanying evaluation will be carried out.

DETAILED DESCRIPTION:
IMPLEMENT is an exploratory, open-label, non-randomized, mixed-methods study. No additional treatments or therapies that can influence the course of the disease are provided to the participating patients. Rather, various implementation strategies will be developed to bring more patients into the existing quality-assures oncological exercise therapy (qOET), to further develop other exercise and sports offers for qOET or to create completely new offers of qOET. The implementation strategies are examined with regard to their degree of effectiveness. The effectiveness is determined by means of a before-and-after comparison (e.g. number of patients in qOET at baseline) and, if applicable, with comparable studies. IMPLEMENT is evaluated using the RE-AIM framework. The aim of the data collection carried out in IMPLEMENT is to provide the necessary data for the evaluation with RE-AIM on the one hand, and to provide information for the development and adaptation of suitable implementation strategies on the other.

Risks to achieving the objectives include the willingness of patients to participate in qOET and the willingness of doctors, therapists and other people working in oncological care to implement the interventions and to expand and adapt their professional activities accordingly. To address these challenges, a mixed-methods approach is used to identify barriers and facilitators. A mixed-methods approach enables a theoretical understanding of the implementation process and provides a more comprehensive picture of the factors relevant to successful implementation than qualitative or exclusively quantitative methods alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer
* Healthcare providers (e.g. Medical Doctors, physiotherapists, nurses, psychologists) involved in the treatment and/or counseling of cancer patients, including aftercare.

Exclusion Criteria (Cancer Patients):

* Psychological and/or physical limitations that do not allow participation in quality-assured sports and exercise therapy (e.g. unstable cardiac arrhythmias)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Increase oncology patients participating in quality-assured exercise therapy | Baseline (M1), one year (M2) and 2 years (M3)
  The primary outcome of the IMPLEMENT project is an increase in the number of oncology patients participating in quality-assured sports and exercise therapy (median 30%). The primary outcome is measured by the RE-AIM (Reach) questionnaire in a semi-structured personal interview three times.

SECONDARY OUTCOMES:
SO1. Adoption/acceptance | Baseline (M1), one year (M2) and 2 years (M3)
  Indicator: Other IMPLEMENT locations or institutions offer quality-assured exercise therapy.
  Indicator: The existing quality-assured exercise therapy service is offered to other oncology patient groups.
  These outcomes are measured using the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) questionnaire in a semi-structured personal interview three times. We report the overall numbers, higher is better.
SO2. Patient-related effectiveness | Baseline (M1), one year (M2) and 2 years (M3)
  Indicator: Proportion of patients who report a positive impact of exercise therapy on their daily lives (increase of 25% over the course of the project).
  Patient-related effectiveness is measured using the quality of life questionnaires (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) for adults and Pediatric Quality of Life Inventory™ Version 4.0. (PedsQL™ 4.0) for children and adolescents. The EORTC QLQ-C30 is a 30 item instrument meant to assess some of the different aspects that define the quality of life of cancer patients. The 23-item PedsQL™ 4.0 measures health-related quality of life (HRQoL) in children and adolescents across multiple dimensions, including physical, emotional, social, and school functioning. Results will be transformed into scores on a 0-100 scale, with higher scores indicating better HRQoL.
SO3. Consistency of implementation | Baseline (M1), one year (M2) and 2 years (M3)
  Indicator: At all IMPLEMENT locations and institutions, a) participation in the standardized IMPLEMENT further education and training program is offered at the IMPLEMENT location in Cologne (face-to-face or online) and b) if the institution offers quality-assured exercise therapy, the standardized further education and training program is taken up by at least 50% of the therapists working in quality-assured exercise therapy.
  Indicator: At all institutions that offer quality-assured exercise therapy, at least 80% of patients are informed about the offer.
  These outcomes are measured using the RE-AIM (Consistency of implementation) questionnaire in a semi-structured personal interview three times. We report proportions, 0-100%, higher is better.
SO4. Maintenance | Baseline (M1), one year (M2) and 2 years (M3)
  Indicator: Quality-assured exercise therapy can be offered beyond the course of the project at all IMPLEMENT locations and institutions that started quality-assured exercise therapy during the course of the project.
  Indicator: Information on financing models (e.g. with health insurance companies) from all IMPLEMENT locations and institutions has been summarized centrally in IMPLEMENT and is included in the recommendations for the sustainable implementation of quality-assured exercise therapy.
  These outcomes are measured using the RE-AIM (Maintenance) questionnaire in a semi-structured personal interview three times. We report proportions, 0-100%, higher is better.

CONTACTS AND LOCATIONS:
Overall Officials: Freerk Baumann, Prof. Dr., Principal Investigator — University of Cologne; Michael Leitzmann, Prof.Dr.Dr., Principal Investigator — University of Regensburg; Hajo Zeeb, Prof. Dr., Principal Investigator — Leibniz Institute for Prevention Research and Epidemiology - BIPS GmbH
Locations (1):
- University Hospital Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No